CLINICAL TRIAL: NCT01258998
Title: Phase II Study of MK-2206 in Patients With Relapsed Lymphoma
Brief Title: Study of Akt Inhibitor MK2206 in Patients With Relapsed Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02890; NCI-2012-02890 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2011-00275; 2010-0261 (Other: M D Anderson Cancer Center); 8728 (Other: CTEP); N01CM00039 (NIH); P30CA016672 (NIH); N01CM62202 (NIH)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; B-cell Adult Acute Lymphoblastic Leukemia; B-cell Chronic Lymphocytic Leukemia; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; T-cell Adult Acute Lymphoblastic Leukemia; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Leukemia, Lymphocytic, Chronic, B-Cell; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — MK 2206

ARMS (1):
- Treatment (Akt inhibitor MK2206) (Experimental): Patients receive Akt inhibitor MK2206 PO once weekly. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt inhibitor MK2206; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Akt inhibitor MK2206 — Given PO
  Other Names: MK2206
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II clinical trial studies how well Akt inhibitor MK2206 works in treating patients with relapsed lymphoma. Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate (ORR) of MK-2206 (Akt inhibitor MK2206) in patients with relapsed/refractory lymphoma.

SECONDARY OBJECTIVES:

I. Assess the progression free survival (PFS) of MK-2206 in patients with relapsed/refractory lymphoma.

II. Assess the safety and tolerability of MK-2206 monotherapy. III. Examine pretreatment phosphorylated v-akt murine thymoma viral oncogene homolog 1 (pAkt) protein expression by immunohistochemistry, and correlate the results with treatment response.

IV. Examine the effect of therapy on serum cytokines and chemokines that regulate the tumor-promoting inflammatory process and/or immunity in patients with relapsed/refractory lymphoma, and correlate the results with treatment response.

OUTLINE:

Patients receive Akt inhibitor MK2206 orally (PO) once weekly. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Hodgkin lymphoma (HL) or non-Hodgkin lymphoma (NHL) (small lymphocytic lymphoma may be included)
* Relapsed or refractory after at least one regimen and with no curative option with conventional therapy
* Bidimensionally measurable disease (at least 2 cm)
* No evidence of cerebral or meningeal involvement by lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Signed informed consent form prior to enrollment
* Women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a women become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately

Exclusion Criteria:

* Burkitt's lymphoma, lymphoblastic lymphoma, chronic lymphocytic leukemia and cutaneous T-cell lymphoma
* Chemotherapy or radiation therapy or other investigational agents within 3 weeks prior to entering the study unless there is clear evidence of progression of disease and toxicity from previous treatment has resolved in which case study entry may be within 1 week of last treatment
* Previous radioimmunotherapy within 12 weeks
* Patients with known immunodeficiency virus (HIV) infection must not have cluster of differentiation (CD)4 cells < 400/mm^3 and who must not have a prior acquired immunodeficiency syndrome (AIDS)-defining diagnosis and cannot be on antiretroviral therapy for HIV
* Known active viral hepatitis
* Any serious active disease or co-morbid condition, which in the opinion of the principal investigator, will interfere with the safety or with compliance with the study
* Absolute neutrophil count < 1.5 x 10^9/L
* Platelets < 75 x 10^9/L
* Total bilirubin > 1.5 x upper limit of normal (ULN) (> 3 x ULN for patients with liver involvement)
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 2.5 x ULN (> 5 x ULN for patients with liver involvement)
* Serum creatinine > 2 x ULN
* Hemoglobin (Hb)A1C > 8%
* Patients receiving any medications or substances that are inhibitors of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP 450 3A4) are ineligible
* Patients with diabetes or in risk for hyperglycemia should not be excluded from trials with MK-2206, but the hyperglycemia should be well controlled on oral agents before the patient enters the trial
* Cardiovascular: baseline Fredericia corrected QT interval (QTcF) > 450 msec (male) or QTcF > 470 msec (female) will exclude patients from entry on study
* Significant heart block or baseline bradycardia < 50 beats per minute (bpm) due to cardiac disease
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Oki, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Oki Y, Fanale M, Romaguera J, Fayad L, Fowler N, Copeland A, Samaniego F, Kwak LW, Neelapu S, Wang M, Feng L, Younes A. Phase II study of an AKT inhibitor MK2206 in patients with relapsed or refractory lymphoma. Br J Haematol. 2015 Nov;171(4):463-70. doi: 10.1111/bjh.13603. Epub 2015 Jul 27. PMID 26213141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 10, 2010 to February 20, 2013. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Akt Inhibitor MK2206: Akt inhibitor MK2206 200 mg orally once a week, repeats every 28 days for up to 12 courses.
Period: Overall Study
Arm/Group | Akt Inhibitor MK2206
Started | 60
Completed | 59
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Akt Inhibitor MK2206): Akt inhibitor MK2206 200 mg orally once a week, repeats every 28 days for up to 12 courses.
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 58 [21 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Complete Response (CR) Disappearance of all evidence of disease(a) FDG-avid or PET positive prior to therapy; mass of any size permitted if PET negative (b) Variably FDG-avid or PET negative; regression to normal size on CT Not palpable, nodules disappeared Infiltrate cleared on repeat biopsy; if indeterminate by morphology, immuno histochemistry should be negative.
  Partial Response (PR) Regression of measurable disease and no new sites, 50% decrease in , sum of the product of the diameters SPD of up to 6 largest dominant masses; no increase in size of other nodes(a) FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site (b) Variably FDG-avid or PET negative; regression on CT, 50% decrease in SPD of nodules (for single nodule in greatest transverse diameter); no increase in size of liver or spleen, Irrelevant if positive prior to therapy; cell type should be specified.
Time Frame: 4 months
Population: Based on intent-to-treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Akt Inhibitor MK2206
Number analyzed (Participants) | 59
Participants
  Complete Response (CR) | 2
  Partial Response (PR) | 6

2. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier method was used. The log-rank test was performed to test the difference in time-to-event distributions between patient groups. Cox proportional hazards model was used to include multiple covariates in the time-to-event analysis.
Time Frame: From treatment start date until the date of first documented progression or date of death from any cause, whichever came first.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Akt Inhibitor MK2206
Number analyzed (Participants) | 59
months | 2.8 [2 to 6]

3. Secondary Outcome: Duration of Response
Description: as for outcome 2
Time Frame: From the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.
Measure: Median (Full Range); unit: months
Arm/Group | Akt Inhibitor MK2206
Number analyzed (Participants) | 59
months | 5.8 [1.8 to 11.6]

4. Secondary Outcome: Overall Survival
Description: Number of surviving participants without disease progression or death for any reason at one year post treatment. Kaplan-Meier method was used.
Time Frame: From the start of treatment to death or 30 days after removal from the study whichever occurs first
Population: PI is not available, therefore, no data is available for reporting in this section due to the overall survival was not an outcome to be measured initially. All efforts were made to retrieve data.
Arm/Group | Akt Inhibitor MK2206
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Change in Cytokine Levels With p Values <0.05
Description: The changes in the cytokine levels from baseline analyzed by Wilcoxon signed rank test. P values < 0.05 were considered statistically significant.
Time Frame: Baseline to up to 30 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Akt Inhibitor MK2206
Number analyzed (Participants) | 36
Participants | 36

6. Secondary Outcome: Number of Participants With Change in Chemokine Levels With p Values <0.05
Description: The changes in the chemokine levels from baseline analyzed by Wilcoxon signed rank test. P values < 0.05 were considered statistically significant.
Time Frame: Baseline to up to 30 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Akt Inhibitor MK2206
Number analyzed (Participants) | 36
Participants | 0

7. Secondary Outcome: Number of Participants With Change in Biomarker Levels With p Values <0.05
Description: as for outcome 5
Time Frame: Baseline to up to 30 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Akt Inhibitor MK2206
Number analyzed (Participants) | 36
Participants | 0

8. Secondary Outcome: Incidence of Adverse Events as Graded by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Toxicity data will be summarized by frequency tables.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Akt Inhibitor MK2206
Number analyzed (Participants) | 59
Participants
  Fatigue | 12
  Anorexia | 4
  Aspartate aminotransferase elevation | 4
  Constipation | 3
  Diarrhea | 4
  Nausea | 9
  Hyperglycemia | 34
  Elevated creatinine | 4
  Conjunctivitis | 4
  Rash | 31
  Dry skin | 4
  Pruritus | 6
  Anemia | 5
  Thrombocytopenia | 15
  Neutropenia | 10
  Lymphopenia | 13

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the time of the first treatment to discontinuation of participant in study, up to 3 years.
Groups:
- Treatment (Akt Inhibitor MK2206): Akt inhibitor MK2206 orally once a week, repeats every 28 days for up to 12 courses.
Arm/Group | Treatment (Akt Inhibitor MK2206)
Serious Adverse Events (participants affected / at risk) | 5/60
Other Adverse Events (participants affected / at risk) | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=60)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=60)
Abdominal pain (Gastrointestinal disorders) | 1 (4)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 1 (8)
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 1 (29)
Allergic rhinitis (Immune system disorders) | 2 (14)
Anemia (Blood and lymphatic system disorders) | 11 (71)
Anorexia (Gastrointestinal disorders) | 1 (9)
Anxiety (Nervous system disorders) | 2 (10)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (3)
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 3 (12)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 (6)
Blurred vision (Eye disorders) | 1 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (3)
Chest wall pain (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Chills (General disorders) | 1 (2)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (2)
Conjunctivitis (Eye disorders) | 1 (5)
Constipation (Gastrointestinal disorders) | 1 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (22)
Creatinine increased (Blood and lymphatic system disorders) | 1 (14)
Dehydration (Gastrointestinal disorders) | 1 (2)
Depression (Nervous system disorders) | 3 (8)
Diarrhea (Gastrointestinal disorders) | 2 (12)
Dizziness (Nervous system disorders) | 1 (5)
Dry eye (Eye disorders) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (7)
Dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (12)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema limbs (Blood and lymphatic system disorders) | 1 (10)
Edema trunk (Blood and lymphatic system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2)
Eye pain (Eye disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Facial pain (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 4 (24)
Fever (General disorders) | 1 (14)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (4)
General disorders and administration site conditions (General disorders) | 2 (4)
Headache (Nervous system disorders) | 1 (10)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (8)
Hyperglycemia (Blood and lymphatic system disorders) | 5 (89)
Hyperkalemia (Blood and lymphatic system disorders) | 2 (14)
Hypernatremia (Blood and lymphatic system disorders) | 1 (4)
Hypertension (Cardiac disorders) | 4 (8)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypertriglyceridemia (Blood and lymphatic system disorders) | 1 (1)
Hyperuricemia (Blood and lymphatic system disorders) | 1 (4)
Hypoalbuminemia (Blood and lymphatic system disorders) | 3 (16)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (9)
Hypoglycemia (Blood and lymphatic system disorders) | 2 (4)
Hypokalemia (Blood and lymphatic system disorders) | 1 (6)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (16)
Hyponatremia (Blood and lymphatic system disorders) | 1 (5)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (16)
Hypotension (Cardiac disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (5)
Infections and infestations (Infections and infestations) | 1 (4)
Insomnia (General disorders) | 1 (6)
Investigations (Investigations) | 1 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Lethargy (General disorders) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 3 (13)
Lymphedema (Blood and lymphatic system disorders) | 1 (2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (59)
Malaise (General disorders) | 1 (3)
Memory impairment (Nervous system disorders) | 1 (1)
Mucosal infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Nausea (Gastrointestinal disorders) | 1 (15)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Neutrophil count decreased (Blood and lymphatic system disorders) | 3 (19)
Non-cardiac chest pain (Cardiac disorders) | 1 (1)
Pain (General disorders) | 2 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (5)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (15)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 3 (47)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (16)
Psychiatric disorders (Psychiatric disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (59)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 1 (5)
Seizure (Nervous system disorders) | 1 (1)
Sinus bradycardia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (4)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Tinnitus (Ear and labyrinth disorders) | 1 (5)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (11)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3)
Weight loss (General disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Blood and lymphatic system disorders) | 3 (29)
Wrist fracture (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less